CLINICAL TRIAL: NCT06427889
Title: A Superiority Study Comparing Two Pharmaceutical Skin Care Creams Containing Different Humectants with a Non-humectant Containing Skin Care Cream for the Treatment of Xerotic Foot of Persons with Diabetes
Brief Title: Treatment Effects of Two Pharmaceutical Skin Care Creams for Xerotic Feet Among Persons with Diabetes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Tautgirdas Ruzgas, Professor,Biomedical technology, Study director, Malmö University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-500907-27-01
Record Dates: First submitted 2024-05-03; First posted 2024-05-24 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus; Skin and Connective Tissue Diseases
Keywords: Diabetes Mellitus; Dry Skin; Self Care; Dry Feet; Prevention
MeSH Terms: conditions — Diabetes Mellitus; Skin and Connective Tissue Diseases | interventions — Decubal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Canoderm (Experimental): Topical on feet twice a day
  Interventions: Drug: Canoderm
- Oviderm (Experimental): Topical on feet twice a day
  Interventions: Drug: Oviderm
- Decubal (Active Comparator): Topical on feet twice a day
  Interventions: Drug: Decubal

INTERVENTIONS:
Drug: Canoderm — humectant
  Arms: Canoderm
Drug: Oviderm — humectant + antimicrobial
  Arms: Oviderm
Drug: Decubal — Non-humectant
  Arms: Decubal

SUMMARY:
Introduction Diabetic foot-ulcers leads to decreased quality of life, risk of major amputation, and resource demanding health-care. To minimize the risk of developing foot-ulcers, persons with diabetes are given the advice to daily inspect their feet and to apply skincare formulations. However, commercially available skincare products have rarely been developed and evaluated for diabetes foot care specifically. The primary aim of this randomized controlled trial (RCT) is to evaluate the effects in reducing foot xerosis in persons with diabetes without foot-ulcers using two skincare creams containing different humectants (interventions) against a cream base non-humectant (comparator). Secondary outcomes are to evaluate differences on skin barrier integrity, low-molecular weight biomarkers and skin microbiota, microcirculation including transcutaneous oxygen pressure, degree of neuropathy, and HbA1c between intervention-comparator cream. Methods Two-armed double-blind RCT. With 80% power, two-tailed significance of 2.5% in each arm, 39 study persons is needed in each arm, total 78 persons, to be able to prove a reduction of at least one category in the Xerosis Severity Scale with the intervention creams compared to the comparator. In one arm, each participant will treat one foot with one of the intervention creams (Oviderm® or Canoderm®), while the opposite foot will be treated with the comparator cream (Decubal® lipid cream®), twice a day. If needed, participants are enrolled after a wash-out period of two weeks. The participants will undergo examinations at baseline, day 14 and day 28. Discussion This RCT evaluate the potential effects of humectants in skin creams against foot xerosis in persons with diabetes. The outcomes of this trial could have implications on treatment recommendations of foot care and for the prevention of foot ulcer.

ELIGIBILITY:
Inclusion Criteria:

* Persons above 18 years of age diagnosed with diabetes mellitus, both type I and II, with self-experienced dry skin.
* Dry skin on both feet with a Xerosis Severity Scale (XSS) score between two to six. No more than one XSS score in difference between the subjects' feet.
* Ability to understand sufficient Swedish language to complete the necessary forms and understand the procedure of the study.

Exclusion Criteria:

* Known sensibility to any of the ingredients in the products.
* Other diagnosed skin disease on the feet.
* Active lesions on either foot.
* Treatment with local medications, including topical moisturizers or keratolytic agents on the feet, within two weeks before the beginning of the study.
* Potential study subjects judged unable to comply with treatment schedule and study specific information.
* Female of childbearing potential that do not use effective medically accepted contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-11-07 (Estimated); Study Completion 2026-08-07 (Estimated)

PRIMARY OUTCOMES:
Xerosis Severity | 4 weeks
  Change in Xerosis Severity (Scale scores 0 - 6, 6 is the worst)

SECONDARY OUTCOMES:
Transepidermal water loss | 4 weeks
  Trans epidermal water loss (TEWL) (grams per square meter per hour)
Skin resistance | 4 weeks
  Skin resistance in Ohms (Ω)
Skin Capacitance | 4 weeks
  Skin Capacitance in Farads (F)
Skin pH | 4 weeks
  Skin pH (5-8)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Kumlien, Professor, Principal Investigator — Malmo University
Locations (1):
- Malmö University, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ericsson A, Borgstrom K, Kumlien C, Gershater Annersten M, Ruzgas T, Engblom J, Gudmundsson P, Lazer V, Jankovskaja S, Lavant E, Agren-Witteschus S, Bjorklund S, Salim S, Astrom M, Acosta S. Treatment effects of two pharmaceutical skin care creams for xerotic feet among persons with diabetes: Rationale and design of a two-armed double blind randomized controlled trial. Contemp Clin Trials Commun. 2024 Sep 16;42:101372. doi: 10.1016/j.conctc.2024.101372. eCollection 2024 Dec. PMID 39345688